CLINICAL TRIAL: NCT02045355
Title: Effects of Fish or Meat Consumption on Sarcopenia and Mobility in Elderly After Hip Fracture
Brief Title: Effects of Fish or Meat Consumption in Elderly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients to recruite.
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Jutta Dierkes, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013/2004-WP4
Record Dates: First submitted 2014-01-17; First posted 2014-01-24 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Sarcopenia; Hip Fractures
MeSH Terms: conditions — Sarcopenia; Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish intervention (Experimental): The patients will receive one portion of salmon (150 g), one portion of cod (150 g), and two portions of sild (50g each) per week.
  Interventions: Other: Fish intervention
- Meat control group (No Intervention): The control food will be pork and chicken (150 g each) and two portions of cooked ham / liver pate for use in cold meals (50 g each).

INTERVENTIONS:
Other: Fish intervention — The intervention will compare fish intake with a correspondent amount of meat. The basis for the comparison will be the estimated protein intake from fish and meat and should be almost similar both from fish and from meat. To ensure compliance and to add more variety to the diet, different fish types will be included in the intervention group and different meat sources in the control group. The types of fish (and that of meat in the control diet) that will be used will be accurately documented and will be similar for all participants included.
  Arms: Fish intervention

SUMMARY:
Health effects of fish consumption have been demonstrated in epidemiological studies and in controlled intervention studies in a number of different population groups, however, randomized controlled studies on the effect of fish consumption in elderly are sparse. Many studies have focused on n-3 fatty acids instead of fish as a food and therefore, many health effects have only been related to the effect of n- 3 fatty acids. The elderly are a heterogeneous population group and therefore difficult to study. In order to reduce heterogeneity, it is advisable to focus on elderly with specific needs. Elderly who experienced a hip fracture can serve as a model for an advanced ageing process, as these patients typically experience a huge inflammatory response, immobilisation and a reduction in muscle mass. Increased fish intake is believed to have effects towards inflammation and a reduction in muscle mass. Therefore, we want to test whether increased fish intake can have positive health effects in elderly who experienced a hip fracture.

Main hypothesis:

Increased fish intake (salmon, cod, pelagic fish), in comparison to meat, will increase mobility, muscle strength and mobility in frail elderly.

Objectives

1. To evaluate the health effects of fish consumption in frail elderly The effect of a dietary intervention with fish on mobility, muscle mass and strength in elderly who experienced a hip fracture has not been shown before.
2. To demonstrate the feasibility of dietary intervention in elderly We want to show that a dietary intervention with fish or control meals is feasible in elderly. The meals (4 portions of fish per week or control portions of meat) will be delivered to their homes.

Description of work and role of participants This is a randomized clinical trial (RCT) on the effect of fish consumption on mobility in elderly who experienced a hip fracture. Elderly who experienced a hip fracture but were able to walk without support by a person before the fracture, will receive, after being randomized to two groups, fish or meat to be used in cold or warm meals at 4 days per week for a period of 16 weeks. Measurements will be taken at baseline (when patients have left the rehabilitation center), after 4 weeks and after 16 weeks. Measurements at 4 and 16 weeks after inclusion will be at their homes or in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients >65 years with a first hip fracture who have a reasonable high chance of returning to their homes after rehabilitation,
* with a sufficient cognitive function to understand the objectives of the study
* the ability to go / walk without support of a person prior to the hip fracture.
* the life expectancy should be more than 6 months.
* the ability to use the provided food and willingness to participate
* sign the informed consent.

Exclusion Criteria:

* Patients are excluded who will probably not return to their home but to a nursing home.
* Patients who lack the cognitive function to understand the study objectives
* Patients with a missing informed consent
* Patients with reduced life expectancy of less than 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change in New Mobility Score (NMS) | Baseline and 16 weeks
  The NMS is an easy, reliable tool for the assessment of mobility. It is based on three questions, which are scored with 0 to 3, thus the result will be between 0 and 9 points.

SECONDARY OUTCOMES:
Change of muscle mass | Baseline and 16 weeks
  Measure muscle mass by using Bioelectrical impedance (BIA Anniversary 100)
Change in Vitamin D status | Baseline and 16 weeks
  Measurement of serum 25OHD.
Change of muscle strength | Baseline and 16 weeks
  Hand grip measurement (JAMAR).
Change of self-perceived health | Recruitment and 4 months
  Standardized questionnaire (EuroQol 5D)

OTHER OUTCOMES:
Change in inflammation | Baseline and 16 weeks
  Measurement of C-reactive protein in blood samples
Change of dietary habits | Baseline and 16 weeks
  Assessment of dietary habits using 24 hour recall.
Number of falls during intervention period | 16 weeks
  Weekly assessment of falls in the previous week by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Dierkes, Principal Investigator — Departmente of Clinical Medicine, University of Bergen; Oddrun A Gudbrandsen, Principal Investigator — Department of Clinical Medicine, University of Bergen
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen, Hordaland
  - Haraldsplass Deacon Hospital, Bergen, Hordaland

REFERENCES:
- [Background] Parker MJ, Palmer CR. A new mobility score for predicting mortality after hip fracture. J Bone Joint Surg Br. 1993 Sep;75(5):797-8. doi: 10.1302/0301-620X.75B5.8376443.